CLINICAL TRIAL: NCT04530760
Title: Impact of Intraabdominal Hypertension on Microaspiration Incidence in Cirrhotic Patients
Brief Title: Intraabdominal Hypertension and Occurrence of Microaspiration in Cirrhotics Under Mechanical Ventilation
Acronym: ATOMIC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_75; 2019-A02622-55 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-27; First posted 2020-08-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness; Cirrhosis, Liver
MeSH Terms: conditions — Critical Illness; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- intraabdominal hypertension group: patients with intraabdominal hypertension defined as intravesical pressure more than 12 mmHg
- control group: patients with no intraabdominal hypertension

SUMMARY:
The study aims to demonstrate the relationship between intra-abdominal hypertension (IAH) and abundant microaspirations in mechanically ventilated cirrhotic.

DETAILED DESCRIPTION:
Intra-abdominal pressure monitoring will be performed using intra-vesical pressure every 8 hour in the first 2 days of mechanical ventilation.

Micro aspiration is defined by pepsin or amylase positivity in trachea suction. Two groups will be compared : one with IAH , one without IAH.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* Cirrhosis
* intubation and mechanical ventilation

Exclusion Criteria:

* pregnancy
* oliguric patients
* impossibility to measure intravesical pressure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cirrhotic patients receiving invasive mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 226 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
abundant microaspiration | 48 hours after inclusion
  presence of pepsin or alpha amylase at significant level in at least 30% of tracheal aspirates

SECONDARY OUTCOMES:
Mortality | from ICU admission until day 28
  number of death
Incidence of ventilator associated pneumonia (VAP) | from intubation until day 28 or extubation
  percentage of patients with VAP
duration of mechanical ventilation | from intubation until day 28 or extubation
  number of days with mechanical ventilation
incidence of patients requiring renal replacement therapy | from ICU admission until Day 28 or ICu discharge, whichever came first
  percentage of patients with renal replacement treatment
incidence of cirrhosis related complications | from ICU admission until Day 28 or ICU discharge, whichever came first
  percentage of patients with cirrhosis related complications

CONTACTS AND LOCATIONS:
Overall Officials: Saad Nseir, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (2):
- France (2):
  - Hop Claude Huriez Chu Lille, Lille
  - Hop Salengro - Hopital B, Lille